CLINICAL TRIAL: NCT03569995
Title: Combination of Rituximab and Methotrexate Followed by Rituximab and Cytarabine in Elderly Patients With Primary CNS Lymphoma
Brief Title: [CREMA]Combination of R-M Followed by R-A in Elderly Patients With Primary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Won Seog Kim (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor-Investigator, Won Seog Kim, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-12-103
Record Dates: First submitted 2018-05-07; First posted 2018-06-26 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Primary CNS Lymphoma
MeSH Terms: interventions — Rituximab; Methotrexate; Cytarabine

STUDY DESIGN:
Intervention Model Description: [Induction phase]
  ① After induction therapy (R-M) 2 times, first evaluation
  * Complete, partial response or stable disease-> next step
  * Progressive disease-> eliminated
    ② After Induction therapy (R-M) was added 3 times (total 5 times), 2nd evaluation
  * Complete response -> consolidation therapy progress
  * Partial response or stable disease-> R-M 2 additional administrations
  * Progressive disease-> eliminated
    ③ After Induction therapy (R-M) was added twice (7 times in total), 3rd evaluation
  * Complete, partial response or stable disease-> consolidation therapy
  * Progressive disease-> eliminated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction+Consolidation chemotherapy (Experimental): [Induction phase]
  ① After induction therapy (Rituximab-Methotrexate) 2 times, first evaluation
  * Complete, partial response or stable disease-> next step
  * Progressive disease-> eliminated
    ② After Induction therapy (Rituximab-Methotrexate) was added 3 times (total 5 times), 2nd evaluation
  * Complete response -> consolidation therapy(Rituximab-Cytarabine) progress
  * Partial response or stable disease-> Rituximab-Methotrexate 2 additional administrations
  * Progressive disease-> eliminated
    ③ After Induction therapy (Rituximab-Methotrexate) was added twice (7 times in total), 3rd evaluation
  * Complete, partial response or stable disease-> consolidation therapy(Rituximab-Cytarabine)
  * Progressive disease-> eliminated
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Cytarabine Injection

INTERVENTIONS:
Drug: Rituximab — 500 mg/m2 + 5%DW 500 mL IVF Begin with 50 mg/hr (increase by 50 mg/hr per 30 min until 400 mg/hr is reached)
  Other Names: Truxima Inj
Drug: Methotrexate — 500 mg/m2 + 5%DW 200 mL IV over 15 minutes 3000 mg/m2 + 5%DW 500 mL IVF over 3 hrs Concurrent hydration and subsequent leucovorin rescue is mandatory
  Other Names: Methotrexate Inj
Drug: Cytarabine Injection — 3000 mg/m2 + 5%DW 200 mL IVF over 2 hrs steroid eye drop 0.1%, 2 drops q 6hrs, on days 1-9
  Other Names: Cytarabine

SUMMARY:
This study was conducted to evaluate the 2-year progression free survival rate of elderly patients with primary CNS lymphoma followed by combination of rituximab and methotrexate followed by rituximab and cytarabine.

DETAILED DESCRIPTION:
As described, standard therapy for patients with primary CNS lymphoma is not based on a high level of evidence yet, and studies in elderly patients with this disease are very limited. Based on the Korea National Cancer Incidence Database, it is estimated that about 100 ~ 150 cases of primary central nervous system lymphoma are diagnosed per year in Korea, but there is no analysis through prospective studies. As described previously, MTX monotherapy in elderly patients is relatively safe and does not reduce clinical utility. Although the autologous therapy may consider autologous stem cell transplantation, it is difficult to apply in elderly patients. Brain radiation therapy is not a primary consideration because it may cause neurological sequelae, especially in elderly patients. High-dose cytarabine is a safely administered drug that has been used extensively in clinical studies involving the treatment of elderly patients.Rituximab has not been studied prospectively for medications, doses, and intervals that are expected to play a role in patients with primary CNS lymphoma, as described above, and may be caused by reducing the number of cytotoxic anticancer drugs in elderly patients And to reduce the treatment effect.

Therefore, the authors propose a two-phase study in which R-A induction therapy is performed after R-M induction therapy in elderly patients with primary CNS lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of B-cell non-Hodgkin's lymphoma, exclusively localized in the central nervous system, cranial nerves, and/or eyes
2. No previous treatment; A tumorectomy on diagnostic purpose and/or use of glucocorticoids is allowed
3. Measurable lesion(s)
4. Age ≥ 60 years
5. Unfit patients for high-dose chemotherapy followed by autologous stem cell transplantation
6. Adequate organ functions

   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
   * Platelets ≥ 50 x 109/L
   * Hemoglobin ≥ 8.0 g/dL
   * Serum Creatinine ≤ 1.5 x upper limit normal (ULN)
   * Serum Bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 3 x ULN
7. Patients with adequately controlled HBV, HCV or HIV are allowed. In case of HBV (+), adequate anti-viral prophylaxis should be incorporated. In case of HIV (+), highly active anti-retroviral therapy should be incorporated.
8. Written informed consent
9. ECOG performance scale 0, 1 or 2
10. Life expectancy > 3 months

Exclusion Criteria:

1. T-cell or NK/T cell lymphoma
2. Any evidence of systemic non-Hodgkin's lymphoma as demonstrated by computed tomography scan of the neck, chest, abdomen, and pelvis and bone marrow examinations
3. Young and fit patients who are suitable for high-dose chemotherapy followed by autologous stem cell transplantation
4. Prior radiation therapy on target CNS lesion(s)
5. Concurrent severe or uncontrolled medical conditions, laboratory abnormalities or psychiatric disorders that would preclude the participants in the study by the discretion of attending physicians
6. Metachronous malignancy other than adequately treated basal cell or squamous cell carcinoma of the skin, or CIN of uterine cervix, or prostate cancer that can be observed without treatment
7. Known hypersensitivity to the investigational agent(s)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival rate | the time between the date of treatment start and the date of death due to any cause or date of disease, assessed up to 24 months
  From the end of the last patient's trial, the disease progression will be tracked for up to 2 years, and primary analysis and reporting will be conducted.

SECONDARY OUTCOMES:
progression free survival | 2 years from the date of consent to the date of Progress disease f / u.
  Means the period from the date of consent to the date of disease progression, the time of death, or the last time the disease has not progressed or has confirmed its survival.
overall survival | Time between the start of treatment and the date of death.assessed up to 5 years]
  It measures the time from start of treatment to death.
Frequency of Adverse events classified by each criterion by CTCAE v4.0 | from the date of informed consent signature to 31 days after last drug administration.
  CTCAE v4 (Common Terminology Criteria for Adverse Events v4.0) In the present study, toxicities will be recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Event (CTCAE), version 4.0. Then, the collected Toxicity is classified by CTCAE term and calculated as%, and a lot of AE will be detected.
time to treatment failure | Within 3 years
  Means the period from the date of consent to the date of the onset of the disease or to the discontinuation of treatment for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, M.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu,, South Korea

IPD SHARING:
Plan to Share IPD: No